CLINICAL TRIAL: NCT00906503
Title: Does Ultra Short-term Steroid Therapy Increase the Accuracy of FDG-PET/CT in Evaluation of Pulmonary Nodules?
Brief Title: Fludeoxyglucose F 18-PET/CT Scans in Patients Receiving Ultra Short-Term Dexamethasone For Lung Nodules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000642256; P30CA022453 (NIH); WSU-2008-075
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Nodule
Keywords: pulmonary nodule
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Radioactive Tracers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/Computed Tomography (CT) (Experimental): Four 4 mg dexamethasone tablets by mouth after food 40, 28, 16 and 4 hrs before the scan; Radioactive tracer (18F-FDG), approx. 1 ml (1/5 of a tsp.); Scanned for about 15 minutes for imaging the lungs
  Interventions: Drug: dexamethasone; Procedure: PET/Computed Tomography (CT); Radiation: fludeoxyglucose (18F)

INTERVENTIONS:
Drug: dexamethasone — Four 4 mg dexamethasone tablets by mouth after food 40, 28, 16 and 4 hrs before the scan
  Other Names: Decadron
Procedure: PET/Computed Tomography (CT) — Radioactive tracer (18F-FDG), approx. 1 ml (1/5 of a tsp.); Scanned for about 15 minutes for imaging the lungs
  Other Names: PET Scan
Radiation: fludeoxyglucose (18F) — Radioactive tracer (18F-FDG), approx. 1 ml (1/5 of a tsp.); Scanned for about 15 minutes for imaging the lungs
  Other Names: Radioactive tracer; 18F-FDG

SUMMARY:
RATIONALE: Imaging procedures, such as fludeoxyglucose F 18 (FDG)-PET/CT scan, done before and after steroid therapy may help doctors assess a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase I trial is studying fludeoxyglucose F 18 PET scan performed before and after ultra short-term dexamethasone therapy to see how well it measures changes in nodules in patients with lung nodules.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether ultra short-term steroid therapy (24-48 hours) can be used to increase the accuracy of fludeoxyglucose F 18 positron emission tomography/computed tomography (FDG-PET/CT) imaging in categorizing nodules in patients with pulmonary nodules.
* To calculate the overall sensitivity and specificity of the nodules group, based on FDG uptake, for predicting malignancy.
* To gather effect-size estimates that will be used to improve the quality of a larger follow-up study.

OUTLINE: Patients receive oral dexamethasone at 40, 28, 16, and 4 hours before imaging. Patients undergo fludeoxyglucose F 18 (FDG)-positron emission tomography/computed tomography (PET/CT) imaging at baseline and upon completion of steroid therapy.

After completion of study therapy, patients are followed for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presence of ≥ 1 measurable pulmonary nodule (1.0-3.0 cm) suggestive of malignancy or chronic inflammatory process on positron emission tomography (PET) scan
* No lesions consistent with malignancy or inflammation according to history, PET findings, or biopsy
* Baseline scan average time between injection and start of scan within 50-70 min

  * Mean liver standardized uptake value (SUV) of baseline scan normal
  * No sign of significant partial paravenous tracer administration in the images of baseline scan
* No lung nodule(s) suggestive of lymphoma
* No lung lesions suggestive of tuberculosis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Blood glucose levels ≤ 150 mg/100 mL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to tolerate PET/CT imaging
* No history of diabetes
* No poorly controlled hypertension
* No prior malignancy other than basal cell or squamous cell carcinoma of the skin, carcinoma in situ, or other cancer from which the participant has been disease free for < 3 years

  * No active malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

* More than 5 years since prior chemotherapy or radiotherapy
* No concurrent steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Majid Khalaf, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET/Computed Tomography (CT)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PET/Computed Tomography (CT)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Ultra Short-term Steroid Therapy to Increase the Accuracy of FDG-PET/CT Imaging
Description: The blood glucose of all patients will be checked by accu-check before the injection of 18F-FDG. The acceptable blood glucose level will be ≤120 mg/dl. Any participant experienced elevated fasting blood glucose of more than 120 mg/dl after steroid therapy, he /she will be asked to come back to the PET center within 48 hours to check the blood glucose level. If the blood glucose level did not decline to baseline level, the participant will be asked to follow with his/her family doctor for management. Participants with history of systemic hypertension will be monitored for increased blood pressure. After 50-to-70 minutes period for FDG incorporation into presumed lesions, patient will under go a limited 18F-FDG PET/CT for the area of the interest (1-2 bed positions). PET imaging will be performed using a GE Discovery STE PET/CT system (GE Medical Systems, Milwaukee, WI).
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: gm/ml
Arm/Group | PET/Computed Tomography (CT)
Number analyzed (Participants) | 9
gm/ml
  Malignant nodules | 3.97 (3.81)
  Benign nodules | 4.27 (2.80)
Statistical Analysis 1: Comparison: PET/Computed Tomography (CT); Test type: Superiority or Other; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.06 to 31.1], Standard Deviation 1.6

ADVERSE EVENTS:
Arm/Group | PET/Computed Tomography (CT)
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No